CLINICAL TRIAL: NCT00711243
Title: A Phase I/II Study of Taxotere, Oxaliplatin, and 5- Fluorouracil
Brief Title: Docetaxel, Oxaliplatin, and Fluorouracil in Treating Patients With Metastatic or Unresectable Stomach Cancer, Gastroesophageal Junction Cancer, or Other Solid Tumor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 04I2; P30CA060553 (NIH); NU-0412; SANOFI - AVENTIS-NU0412; NU-948-006; STU00006778 (Other: Northwestern University IRB)
Record Dates: First submitted 2008-07-05; First posted 2008-07-08 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-10

CONDITIONS: Gastric Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; adenocarcinoma of the stomach; stage III gastric cancer; stage IV gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1a (Experimental): Docetaxel 25 mg/m2 + oxaliplatin 85 mg/m2 + 5-Fluorouracil 2.4 gm/m2
  Interventions: Drug: docetaxel; Drug: fluorouracil; Drug: oxaliplatin
- Cohort 2a (Experimental): Docetaxel 30 mg/m2 + oxaliplatin 85 mg/m2 + 5-Fluorouracil 2.4 gm/m2
  Interventions: Drug: docetaxel; Drug: fluorouracil; Drug: oxaliplatin
- Cohort 3a (Experimental): Docetaxel 40 mg/m2 + oxaliplatin 85 mg/m2 + 5-Fluorouracil 2.4 gm/m2
  Interventions: Drug: docetaxel; Drug: fluorouracil; Drug: oxaliplatin
- Cohort 4a (Experimental): Docetaxel 50 mg/m2 + oxaliplatin 85 mg/m2 + 5-Fluorouracil 2.4 gm/m2
  Interventions: Drug: docetaxel; Drug: fluorouracil; Drug: oxaliplatin
- Cohort 5a (Experimental): Docetaxel 60 mg/m2 + oxaliplatin 85 mg/m2 + 5-Fluorouracil 2.4 gm/m2
  Interventions: Drug: docetaxel; Drug: fluorouracil; Drug: oxaliplatin

INTERVENTIONS:
Drug: docetaxel — Docetaxel at the dose indicated by the patient cohort, administered intravenously in 5% dextrose over 1 hour on day 1 of each cycle.
Drug: fluorouracil — Intravenous infusion at 85 mg/m2 continuously over 46 hours beginning each cycle after docetaxel administration.
Drug: oxaliplatin — Oxaliplatin 2.4 gm/m2 administered intravenously in 5% dextrose over 2 hours each cycle beginning immediately following docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, oxaliplatin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of docetaxel when given with oxaliplatin and fluorouracil and to see how well they work in treating patients with metastatic or unresectable stomach cancer, gastroesophageal junction cancer, or other solid tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish the maximum tolerated dose of docetaxel when administered with oxaliplatin and fluorouracil in patients with metastatic or unresectable solid tumors. (Phase I)
* To determine the response rate in patients with metastatic or unresectable adenocarcinoma of the stomach or gastroesophageal junction treated with this regimen. (Phase II)

Secondary

* To determine the dose limiting toxicity of this regimen in these patients.
* To evaluate the frequency of CYP3A4, CYP3A5, and MDR polymorphisms and their impact on toxicity of docetaxel.
* To evaluate the frequency of XRCC1 and ERCC2 polymorphisms and their impact on the toxicity of oxaliplatin.
* To evaluate the frequency of DPD and TSER polymorphisms and their impact on the toxicity of fluorouracil.
* To characterize the toxicity profile of this regimen in these patients.

OUTLINE: This is a dose-escalation study of docetaxel.

Patients receive docetaxel IV over 1 hour and oxaliplatin IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment repeats every 14 days for at least 2 courses in the absence of disease progression, symptomatic tumor progression, or unacceptable toxicity.

Patients undergo blood sample collection periodically for pharmacokinetic and pharmacogenomic correlative studies. Plasma concentrations of docetaxel are analyzed by reverse-phase high performance liquid chromatography and tandem mass spectrometry. Polymorphisms in CYP3A4/5, MDR, and other genes are analyzed by PCR.

After completion of study therapy, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 73 patients (30 for phase I and 43 for phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic or surgically unresectable solid tumor meeting 1 of the following criteria:

  * Any solid tumor (Phase I)
  * Adenocarcinoma of the stomach or gastroesophageal junction (Phase II)
* Unidimensionally measurable disease by CT scan or MRI
* No uncontrolled brain metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin normal
* Meets 1 of the following criteria:

  * Alkaline phosphatase (AP) normal AND AST or ALT ≤ 5 times ULN
  * AP ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST or ALT normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study therapy
* No preexisting neuropathy
* No concurrent uncontrolled illness or other condition that would preclude study compliance
* No history of severe hypersensitivity reaction to docetaxel or to other drugs formulated with polysorbate 80
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in this study

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* More than 4 weeks since prior therapy (Phase I)
* No prior oxaliplatin or taxanes (Phase I)
* More than 4 weeks since prior radiotherapy (Phase I)
* No more than two prior therapies for metastatic disease (Phase I)
* No prior therapy for metastatic disease (Phase II)
* At least 6 months since prior adjuvant therapy (given prior to the occurrence of metastatic disease) (Phase II)
* Prior fluorouracil and concurrent radiotherapy for palliation of the primary tumor allowed provided metastatic disease is present outside the radiotherapy field (Phase II)
* No prior radiotherapy to ≥ 30% of bone marrow
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2005-04-20 (Actual); Primary Completion 2008-12-15 (Actual); Study Completion 2011-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Mulcahy, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Rosenberg AJ, Rademaker A, Hochster HS, Ryan T, Hensing T, Shankaran V, Baddi L, Mahalingam D, Mulcahy MF, Benson AB 3rd. Docetaxel, Oxaliplatin, and 5-Fluorouracil (DOF) in Metastatic and Unresectable Gastric/Gastroesophageal Junction Adenocarcinoma: A Phase II Study with Long-Term Follow-Up. Oncologist. 2019 Aug;24(8):1039-e642. doi: 10.1634/theoncologist.2019-0330. Epub 2019 May 28. PMID 31138725

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on March 3, 2005 and the first patient was enrolled April 20 2005. Accrual goal of approximately 50 for the phase I and phase II portion. Accrual for phase I was suspended on February 13 2006 reopened with phase II accrual on February 16, 2006. The study was closed permanently on July 23, 2008.
Pre-assignment Details: Phase I was opened to all solid tumor cancers and phase II was opened to stomach/gastro-esophageal junction cancer only.
Groups:
- Phase II: Docetaxel 50 mg/m2 + oxaliplatin 85 mg/m2 + 5-Fluorouracil 2.4 gm/m2
  docetaxel: Docetaxel at the dose indicated by the patient cohort, administered intravenously in 5% dextrose over 1 hour on day 1 of each cycle.
  fluorouracil: Intravenous infusion at 85 mg/m2 continuously over 46 hours beginning each cycle after docetaxel administration.
  oxaliplatin: Oxaliplatin 2.4 gm/m2 administered intravenously in 5% dextrose over 2 hours each cycle beginning immediately following docetaxel
Period: Registed and Started Treatment
Arm/Group | Cohort 1a | Cohort 2a | Cohort 3a | Cohort 4a | Cohort 5a | Phase II
Started | 3 | 3 | 3 | 3 | 3 | 44
Registered to Study | 3 | 3 | 3 | 3 | 3 | 44
Started Treatment | 3 | 3 | 3 | 3 | 3 | 43
Completed | 3 | 3 | 3 | 3 | 3 | 43
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Period: Reached First Response/4 Cycles
Arm/Group | Cohort 1a | Cohort 2a | Cohort 3a | Cohort 4a | Cohort 5a | Phase II
Started | 3 | 3 | 3 | 3 | 3 | 43
Completed | 3 | 3 | 3 | 2 | 3 | 41
Not Completed | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Progressive disease | 0 | 0 | 0 | 1 | 0 | 0
Period: Treated Cycle 5 After First Response
Arm/Group | Cohort 1a | Cohort 2a | Cohort 3a | Cohort 4a | Cohort 5a | Phase II
Started | 3 | 3 | 3 | 2 | 3 | 41
Completed | 2 | 1 | 3 | 2 | 2 | 37
Not Completed | 1 | 2 | 0 | 0 | 1 | 4
Not completed — Progressive disease | 1 | 2 | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Decline in performance status | 0 | 0 | 0 | 0 | 0 | 1
Period: Follow up Every 3 Months Until Death
Arm/Group | Cohort 1a | Cohort 2a | Cohort 3a | Cohort 4a | Cohort 5a | Phase II
Started (All patients that are treated on study go into follow up) | 3 | 3 | 3 | 3 | 3 | 39 (4 patients died whilst on study and 1 patient did not get treated on study)
Completed | 3 | 3 | 3 | 3 | 3 | 37
Not Completed | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1a | Cohort 2a | Cohort 3a | Cohort 4a | Cohort 5a | Phase II | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 44 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 1 | 0 | 1 | 28 | 35
  >=65 years | 1 | 0 | 2 | 3 | 2 | 16 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 1 | 2 | 14 | 22
  Male | 1 | 2 | 1 | 2 | 1 | 30 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 3 | 4
  Not Hispanic or Latino | 3 | 2 | 2 | 3 | 3 | 36 | 49
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 8 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 0 | 6 | 8
  White | 2 | 2 | 2 | 3 | 3 | 30 | 42
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 3 | 3 | 3 | 44 | 59

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Docetaxel When Given in Combination With Oxaliplatin and Fluorouracil (Phase I)
Description: The MTD will be determined using a 3+3 dose escalating design. There will be 5 dose cohorts:
  Cohort 1a 25mg/m2 Cohort 2a 30mg/m2 Cohort 3a 40 mg/m2 Cohort 4a 50 mg/m2 Cohort 5a 60 mg/m2
  3 patients will be enrolled at dose of 25mg/m2 docetaxel. If no dose limiting toxicities (DLTs) are seen then dose will be escalated to next cohort and 3 patients will be treated at that dose level. If a DLT is seen at any dose, then 3 more patients will be enrolled at that dose level. If 1 patient out of 6, experience a DLT then MTD will be determined to be at this dose level. If 2 or more DLTs are seen in first 3 patients at that dose, then MTD will be one dose lower to the level where the DLTs were experienced. Dose of docetaxel will be escalated by use of cohorts until the MTD for phase II is determined.
  DLTs were defined using the National Cancer Institute Common Toxicity Criteria Version 3.0
Time Frame: After completion of 1 cycle of therapy (1 cycle = 14 days)
Population: Dose of docetaxel was escalated up through 5 cohorts.
Measure: Number; unit: mg/m2
Groups:
- Phase I: Docetaxel + oxaliplatin 85 mg/m2 + 5-Fluorouracil 2.4 gm/m2
  docetaxel: Docetaxel at the dose indicated by the patient cohort, administered intravenously in 5% dextrose over 1 hour on day 1 of each cycle. Dose for cohorts is as follows: Cohort 1a = Docetaxel 25mg/m2 Cohort 2a = Docetaxel 30mg/m2 Cohort 3a = Docetaxel 40mg/m2 Cohort 4a = Docetaxel 50mg/m2 Cohort 5a = Docetaxel 60mg/m2
  fluorouracil: Intravenous infusion at 85 mg/m2 continuously over 46 hours beginning each cycle after docetaxel administration.
  oxaliplatin: Oxaliplatin 2.4 gm/m2 administered intravenously in 5% dextrose over 2 hours each cycle beginning immediately following docetaxel
Arm/Group | Phase I
Number analyzed (Participants) | 15
mg/m2 | 50

2. Primary Outcome: Response Rate in Patients With Adenocarcinoma of the Stomach or Gastroesophageal Junction (Phase II)
Description: Overall Response Rate (ORR) is defined as Complete Response (CR) plus Partial Response (PR) and will be measured per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT scan.
  Complete Response (CR) - Disappearance of all target lesions. Partial Response (PR), >=30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum.
  Stable Disease, neither sufficient shrinkage to qualify for Partial disease nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD while on study.
  Progressive Disease - <=20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: After 4 cycles of therapy (1 cycle = 14 days)
Population: One patient that was registered to phase II did not get treated on study and was therefore not evaluable. Two patients did not reach first response at 4 cycles and therefore were not evaluable.
Measure: Number; unit: percentage of patients
Groups:
- Phase II: Docetaxel 50mg/m2 + oxaliplatin 85 mg/m2 + 5-Fluorouracil 2.4 gm/m2
  Docetaxel: Docetaxel at the dose indicated by the patient cohort, administered intravenously in 5% dextrose over 1 hour on day 1 of each cycle.
  Fluorouracil: Intravenous infusion at 85 mg/m2 continuously over 46 hours beginning each cycle after docetaxel administration.
  Oxaliplatin: Oxaliplatin 2.4 gm/m2 administered intravenously in 5% dextrose over 2 hours each cycle beginning immediately following docetaxel
Arm/Group | Phase II
Number analyzed (Participants) | 41
percentage of patients | 73.2

3. Secondary Outcome: Dose-limiting Toxicity of Docetaxel When Given in Combination With Oxaliplatin and Fluorouracil
Description: Dose limiting toxicities (DLT) will be graded according to National Cancer Institute's Common Toxicity Criteria for adverse events version 3.0 (CTCAE v3.0) except for neurosensory. The occurrence of any of the following during the 1st cycle, seen in more than one patient, will constitute a DLT.
  Grade 3 non-hematologic toxicity(except alopecia) Grade 4 thrombocytopenia, not recovered to platelet count of >75,000/ul by day 15.
  Grade 4 neutropenia, not recovered to count of >1,500/ul by day 15. Grade 4 neutropenia with fever or infection. Grade 2 neurologic-sensory toxicity not recovered to grade 1 or better by day 15
Time Frame: After 1 cycle of therapy (1 cycle = 14 days)
Population: 15 patients enrolled in 5 dose escalating cohorts were monitored for DLTs in the phase I part of the study.
Measure: Number; unit: participants
Arm/Group | Cohort 1a | Cohort 2a | Cohort 3a | Cohort 4a | Cohort 5a
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
participants
  Fatigue | 0 | 0 | 0 | 0 | 2
  Diarrhea | 0 | 0 | 0 | 0 | 2

4. Secondary Outcome: Frequency of CYP3A4, CYP3A5, and MDR Polymorphisms and Their Impact on Docetaxel Toxicity
Time Frame: Blood sample cycle 1 day 1 and toxicity on day 1 of each cycle
Population: Data not collected.
Groups:
- Phase I and Phase II: Docetaxel (between 25 mg/m2 and 60mg/m2) + oxaliplatin 85 mg/m2 + 5-Fluorouracil 2.4 gm/m2
  docetaxel: Docetaxel at the dose indicated by the patient cohort, administered intravenously in 5% dextrose over 1 hour on day 1 of each cycle.
  fluorouracil: Intravenous infusion at 85 mg/m2 continuously over 46 hours beginning each cycle after docetaxel administration.
  oxaliplatin: Oxaliplatin 2.4 gm/m2 administered intravenously in 5% dextrose over 2 hours each cycle beginning immediately following docetaxel
Arm/Group | Phase I and Phase II
Number analyzed (Participants) | 0

5. Secondary Outcome: Frequency of XRCC1 and ERCC2 Polymorphisms and Their Impact on Oxaliplatin Toxicity
Time Frame: Blood sample cycle 1 day 1 and toxicity on day 1 of each cycle
Population: Data not collected.
Arm/Group | Phase I and Phase II
Number analyzed (Participants) | 0

6. Secondary Outcome: Frequency of DPD and TSER Polymorphisms and Their Impact on Fluorouracil Toxicity
Time Frame: Blood sample cycle 1 day 1 and toxicity on day 1 of each cycle
Population: Data not collected.
Arm/Group | Phase I and Phase II
Number analyzed (Participants) | 0

7. Secondary Outcome: Toxicity Profile
Description: Toxicity data will be collected on day 1 of every 14 day cycle during treatment according to the National Cancer Institute's Common Toxicity Criteria for adverse events (AE) version 3.0 (CTCAE v3.0). For patients that experience multiple grades of the same AE that is determined to be at least possibly related to at least one study drug, only highest grade will be collected. In general AEs will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: Day 1 of each cycle of therapy with 1 cycle =14 days until disease progression for up to a maximum of 34 cycles and 30 days after last treatment
Population: Data collected and analyzed for patients enrolled in the phase II of the study only.1 Patient did not receive treatment on study and was not evaluable. For each patient that experienced the toxicity, highest grade for that patient is recorded. Grades ranging between 1-5 were collected and are represented below.
Measure: Number; unit: participants
Arm/Group | Phase II
Number analyzed (Participants) | 43
participants
  Neutropenia | 23
  Leukopenia | 31
  Lymphopenia | 15
  Anemia | 30
  Thrombocytopenia | 13
  Fatigue | 36
  Vomiting | 22
  Dehydration | 5
  Infection | 4
  Nausea | 31
  Pain | 5
  Allergy | 4
  Transaminitis | 7
  Rash | 3
  Weight loss | 6
  Anorexia | 13
  Fever | 4
  Hypertension | 2
  Hyperglycemia | 3
  Diarrhea | 22
  Constipation | 10
  Mucositis | 14
  Neuro-sens | 30
  Neuro-motor | 2
  Nail changes | 2
  Alopecia | 6
  Skin | 6
  Hemorrhage | 5
  Altered taste | 6
  Edema | 2
  Abdominal distension | 2
  Shortness of breath | 6

8. Post Hoc Outcome: Median Overall Survival (OS)
Description: Median Overall Survival (OS)
Time Frame: From first day of treatment until death from any cause measured, assessed up to 4 years
Population: Patients enrolled in phase II portion of the study were evaluable for OS. One patient in phase II was registered to the study but did not receive treatment and was not evaluable for OS. Two patients did not have death dates and were censored for the last known time to be living.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II
Number analyzed (Participants) | 43
Months | 10.3 [8.1 to 15.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 4 year period across the study.
Description: Adverse events were collected in systematic assessment every two weeks during patient visit. For each patient the highest grade of clinically significant adverse events were collected only.
Groups:
- Cohort 3a: Docetaxel 40 mg/m2+ oxaliplatin 85 mg/m2 + 5-Fluorouracil 2.4 gm/m2
  docetaxel: Docetaxel at the dose indicated by the patient cohort, administered intravenously in 5% dextrose over 1 hour on day 1 of each cycle.
  fluorouracil: Intravenous infusion at 85 mg/m2 continuously over 46 hours beginning each cycle after docetaxel administration.
  oxaliplatin: Oxaliplatin 2.4 gm/m2 administered intravenously in 5% dextrose over 2 hours each cycle beginning immediately following docetaxel
Arm/Group | Cohort 1a | Cohort 2a | Cohort 3a | Cohort 4a | Cohort 5a | Phase II
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 41/43
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 0/3 | 2/3 | 11/43
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a (N=3) | Cohort 2a (N=3) | Cohort 3a (N=3) | Cohort 4a (N=3) | Cohort 5a (N=3) | Phase II (N=43)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Resulted in death
GI bleed (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Resulted in death
Death (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 1 — Reason unknown
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea and vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Speech impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rectal bleeding (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Brain metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 — Found as a result of a seizure
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pleural effusions (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a (N=3) | Cohort 2a (N=3) | Cohort 3a (N=3) | Cohort 4a (N=3) | Cohort 5a (N=3) | Phase II (N=43)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 2 | 1 | 23
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 3 | 3 | 31
Sensory neuropathy (Nervous system disorders) | 1 | 2 | 2 | 2 | 2 | 30
Lymphopenia (Blood and lymphatic system disorders) | 3 | 1 | 3 | 1 | 0 | 15
Diarrhea (Gastrointestinal disorders) | 1 | 3 | 3 | 3 | 2 | 22
Mucositis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 14
Fatigue (General disorders) | 2 | 2 | 3 | 3 | 3 | 36
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 2 | 1 | 2 | 30
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 2 | 1 | 22
Dehydration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 5
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 0 | 1 | 13
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 3 | 1 | 31
Pain (General disorders) | 2 | 1 | 1 | 2 | 2 | 5
Allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 4
Transaminitis (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 7
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 3
Weight loss (General disorders) | 0 | 0 | 1 | 0 | 1 | 6
Anorexia (Gastrointestinal disorders) | 0 | 2 | 3 | 1 | 0 | 13
Fever (General disorders) | 1 | 1 | 0 | 0 | 1 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 10
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1
Albumin, serum low (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0 | 0 | 1
Motor Neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 2 | 6
Skin (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 6
Hemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1 | 5
Altered taste (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 6
Edema (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0 | 2
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 6
Creatinine, Serum high (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Auditory (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
GI distention (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Weight loss (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nose bleed (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Speech (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
GI Bleed (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes